CLINICAL TRIAL: NCT05938777
Title: Efficacy of The Transtheoretical Model of Change in Enhancing High School Female Students' Readiness to Engage in Regular Physical Exercise: A Randomized Controlled Trial
Brief Title: Non-Stage-Matched Intervention to Enhance High School Female Students' Readiness to Engage in Regular Physical Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mohammed Baqer Habeeb Abd Ali, Faculty member, University of Baghdad
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: NSM Regular Physical Exercise
Record Dates: First submitted 2023-06-29; First posted 2023-07-10 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Engaging in Regular Physical Exercise
Keywords: Health Behavior; Regular Physical Exercise; High School Female Students; Transtheoretical Model of Change
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Masking Description: The study participants will be masked from the proposed intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-Stage-Matched Intervention (Experimental): The proposed arm would be non-Stage-matched that involves using different Processes of Change as strategies to enhance engaging in regular physical exercise.
  Interventions: Behavioral: Non-Stage-Matched Intervention

INTERVENTIONS:
Behavioral: Non-Stage-Matched Intervention — The proposed intervention will be non-Stage-Matched that uses different Processes of Change as strategies to change the physical exercise behavior.

SUMMARY:
A non-stage-matched intervention based on the Transtheoretical Model of Change

DETAILED DESCRIPTION:
The proposed intervention would be non-stage-matched intervention based on the Transtheoretical Model of Change.

The study sample would include high school female students (72 for the study group and 72 for the control group). The study participants will be randomly allocated and assigned into each of the study and control groups.

Participants will go through pretest, intervention, posttest 1, and posttest 2. There will be a 12-2eeks interval between the intervention and each of posttest 1 and posttest 2.

ELIGIBILITY:
Inclusion Criteria:

* High school female students who do not experience any physical disability

Exclusion Criteria:

* High school female students who experience any physical disability

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — High school female students will be involved in this study.
Enrollment: 144 (Estimated)
Dates: Start 2024-03-24 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Stages of Change Scale for Regular Physical Exercise | 6 months
  Stages of Change Scale for Regular Physical Exercise

IPD SHARING:
Plan to Share IPD: Undecided